CLINICAL TRIAL: NCT01638468
Title: Pulmonary Embolism Removal With the AngioJet 6F Ultra SystEm (PERFUSE)
Brief Title: Multicenter, Nonrandomized, Prospective Study of Pulmonary Embolism Removal With the AngioJet 6F Ultra System
Acronym: PERFUSE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PERFUSE
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Acute Pulmonary Embolism; Sub-massive Pulmonary Embolism; Massive Pulmonary Embolism; Pulmonary Thromboembolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AngioJet Ultra PE Thrombectomy System (Experimental): Patients are treated with the AngioJet Ultra PE Thrombectomy System
  Interventions: Device: AngioJet Ultra PE Thrombectomy System

INTERVENTIONS:
Device: AngioJet Ultra PE Thrombectomy System — Thrombectomy with or without lytic delivery using the AngioJet Ultra PE Thrombectomy System
  Other Names: AngioJet

SUMMARY:
The purpose of this European Post Market Follow-up Plan is designed to evaluate the safety, efficacy, adverse events and any new information that may surface regarding the use of the AngioJet Ultra PE Thrombectomy Catheter System in patients with thrombus in the main pulmonary and lobar arteries ≥ 6mm in diameter.

DETAILED DESCRIPTION:
Despite advances in prophylaxis, diagnostic modalities, and therapeutic options, pulmonary embolism remains a commonly under diagnosed and lethal entity. In the United States approximately 150,000 patients per year are diagnosed with acute pulmonary embolisms. Many additional deaths occur each year in the United States as a result of undiagnosed massive pulmonary embolisms. Taking these patients into account, it is thought that up to 600,000 patients develop a pulmonary embolism annually in this country. In patients with acute pulmonary embolism, the most common cause of early death is right ventricular failure.

In addition to anticoagulation therapy, several reperfusion therapies are being used to reverse right ventricular failure: systemic thrombolysis, surgical embolectomy, and catheter based therapy. Given the drawbacks of systemic thrombolytic therapy or surgical embolectomy, percutaneous catheter treatment is a reasonable alternative for patients with contraindications to systemic thrombolytic therapy or surgery. Current international consensus guidelines support the use of catheter interventions for selected pulmonary embolism patients at increased risk of adverse clinical outcomes.

The AngioJet Ultra PE Thrombectomy catheter introduces a pressurized high velocity saline stream through a catheter tip so that the clot within a blood vessel is trapped, broken into small pieces and aspirated from the body.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic pulmonary embolism patients >18 years
2. Availability of a baseline contrast-enhanced chest computed tomogram or conventional pulmonary angiogram with evidence of pulmonary embolus in at least one main or lobar pulmonary artery ≥ 6mm in diameter
3. Availability of a baseline transthoracic echocardiogram with sufficient image quality permitting the measurement of right ventricular (RV) and left ventricular (LV) dimensions in the apical or subcostal four-chamber view
4. Echocardiographic evidence of right ventricular dilatation with a subannular RV/LV ratio ≥ 0.9 from the apical or subcostal four-chamber view
5. Appropriate informed consent was obtained from the patient or legal representative

Exclusion Criteria:

1. Patient has underwent Cardiopulmonary Resuscitation (CPR) in the last 48 hours
2. Patient is participating in any other clinical study
3. Pregnancy, lactation or parturition within the previous 30 days (positive pregnancy test, women of childbearing age must be tested or use a medically accepted method of birth control)
4. Inability to comply with study Follow-up assessments (e.g. due to geographic)
5. Previous enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nils Kucher, Prof Dr Med, Principal Investigator — University of Bern
Locations (7):
- Universitätsklinikum Münster, Münster, Germany
- Italy (4):
  - EO Ospedali Galliera - Genova, Genova
  - Universita Federico II di Napoli, Napoli
  - Ospedale S. Maria Delle Croci, Ravenna
  - Ospedale Sant' Anna Di Como, San Fermo della Battaglia
- Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia, Portugal
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AngioJet Ultra PE Thrombectomy System
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AngioJet Ultra PE Thrombectomy System
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Number; unit: participants]
  Italy | 4
  Switzerland | 1
  Portugal | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 28.33 (4.43)
Height [Mean (Standard Deviation); unit: cm] | 170.0 (12.6)
Weight [Mean (Standard Deviation); unit: kg] | 82.6 (19.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Right Ventricular (RV) to Left Ventricular (LV) Ratio at 24 - 48 Hours as Measured by Echocardiography
Description: The change in the subannular end-diastolic RV/LV ratio at 24-48 hrs following thrombectomy compared to baseline measurements as assessed by an independent core lab analysis. RV and LV values will be measured by echocardiography, a technique utilizing ultrasound waves to assess heart activity.
Time Frame: Baseline to 24-48 hours
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AngioJet Ultra PE Thrombectomy System
Number analyzed (Participants) | 7
ratio | -0.610 (0.125)

2. Secondary Outcome: Technical Success
Description: Percentage of patients with successful placement and operation of the AngioJet catheter in the pulmonary arteries during the index procedure
Time Frame: Index Procedure
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | AngioJet Ultra PE Thrombectomy System
Number analyzed (Participants) | 7
percentage of participants | 100

3. Secondary Outcome: Death - All Cause
Description: Number of participant deaths due to any reason occurring within 3 months of the index procedure.
Time Frame: 3 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | AngioJet Ultra PE Thrombectomy System
Number analyzed (Participants) | 7
participants | 1

4. Secondary Outcome: Death - Cardiac Cause
Description: Number of participant deaths due to cardiac causes occurring within 3 months of the index procedure.
Time Frame: 3 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | AngioJet Ultra PE Thrombectomy System
Number analyzed (Participants) | 7
participants | 0

5. Secondary Outcome: Change in Systolic Pulmonary Arterial Blood Pressure
Description: Change in systolic pulmonary arterial blood pressure at termination of the index procedure as compared to the pre-procedure assessment.
Time Frame: Baseline to Post Index Procedure
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 1 participant was not evaluable.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AngioJet Ultra PE Thrombectomy System
Number analyzed (Participants) | 6
mmHg | -8.3 (11.8)

6. Secondary Outcome: Pulmonary Systolic Arterial Blood Pressure
Description: Pulmonary systolic arterial blood pressure at termination of the index procedure.
Time Frame: Post Index Procedure
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 1 participants were not evaluable.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AngioJet Ultra PE Thrombectomy System
Number analyzed (Participants) | 6
mmHg | 44.2 (11.3)

7. Secondary Outcome: Change in Systemic Systolic Arterial Blood Pressure
Description: Change in systemic systolic arterial blood pressure at termination of the index procedure as compared to the pre-procedure assessment.
Time Frame: Baseline to Post Index Procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AngioJet Ultra PE Thrombectomy System
Number analyzed (Participants) | 7
mmHg | 14.7 (22.1)

8. Secondary Outcome: Systemic Systolic Arterial Blood Pressure
Description: Systemic systolic arterial blood pressure at termination of the index procedure.
Time Frame: Post Index Procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AngioJet Ultra PE Thrombectomy System
Number analyzed (Participants) | 7
mmHg | 136.0 (18.5)

9. Secondary Outcome: Change in Heart Rate
Description: Change in heart rate at termination of the index procedure as compared to the pre-procedure assessment.
Time Frame: Baseline to Post Index Procedure
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 2 participants were not evaluable.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | AngioJet Ultra PE Thrombectomy System
Number analyzed (Participants) | 5
beats per minute | -12.2 (9.4)

10. Secondary Outcome: Vasopressor Support
Description: Percentage of participants receiving vasopressor support during the index procedure. Vasopressor support are medications administered to prevent the narrowing of blood vessels.
Time Frame: Index Procedure
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | AngioJet Ultra PE Thrombectomy System
Number analyzed (Participants) | 7
percentage of participants | 0

11. Secondary Outcome: Procedure Related Adverse Event Rate
Description: Number of procedure related adverse events occurring within 3 months of the index procedure
Time Frame: 3 months
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | AngioJet Ultra PE Thrombectomy System
Number analyzed (Participants) | 7
events | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the index procedure through the 3 month follow up visit.
Arm/Group | AngioJet Ultra PE Thrombectomy System
Serious Adverse Events (participants affected / at risk) | 4/7
Other Adverse Events (participants affected / at risk) | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AngioJet Ultra PE Thrombectomy System (N=7)
Pulmonary Embolism, Re-occurring (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Death (Vascular disorders) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Macrohematuria (presence of blood cells in urine) (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AngioJet Ultra PE Thrombectomy System (N=7)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (bleeding from the nose) (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No